CLINICAL TRIAL: NCT01573234
Title: Efficacy of MySkin Patch for the Healing of Cut Injuries and Abrasions: a Randomised Controlled Trial
Brief Title: Efficacy of MySkin Patch for the Healing of Cut Injuries and Abrasions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Associazione Infermieristica per lo studio delle Lesioni Cutanee (Other)
Collaborators: Artsana S.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AISLeC-003
Record Dates: First submitted 2012-04-02; First posted 2012-04-09 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Wounds and Injuries; Abrasion; Cut Injuries
Keywords: MySkin patch; Hydrogel bandage; Occlusive dressing
MeSH Terms: conditions — Wounds and Injuries | interventions — Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MySkin patch (Experimental): Hydrogel and polyurethane film
  Interventions: Device: MySkin patch
- Traditional Dressing (Active Comparator)
  Interventions: Device: Gauze and Patch

INTERVENTIONS:
Device: MySkin patch — Hydrogel and polyurethane film
  Arms: MySkin patch
Device: Gauze and Patch — Traditional Dressing
  Arms: Traditional Dressing

SUMMARY:
Evaluation of clinical efficacy of My Skin (hydrogel and polyurethane film) plus best practice clinical care in subjects with cut injuries and abrasions with particular regard to: Wound healing (complete reepithelialization) and patient's pain.

In the context of the study will be collected secondary outcomes related to type of lesion and its clinical evolution through the analysis of the items in the scale of the Pressure Sore Status Tool(PSST).

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least an injury cut or abrasion (even if sutured)covered by a dressing of 10x8 cm (80 cm2)
* Injury treated with conventional dressings type gauze and patch
* Patients assisted at the emergency care, or at the outpatient
* Extension of the lesion less than 80 cm2 (including dressings in cm10x8cm)
* Patient age greater than or equal to 18 years
* Patients who have given consent to enrollment in the trial and the processing of personal data
* Patient / lesion that has already been recruited in the study or who have previously passed a period of 10 days (wash-out) of "no treatment" according to the research protocol

Exclusion Criteria:

* A end-stage of disease
* Subjected systemic corticosteroid therapy / radiotherapy / immunosuppressive therapy
* Suspected or known allergic diathesis to the product of medication
* Subjects that do not give consent to data processing
* Dry lesion with necrosis or eschar
* Presence of both local and systemic infection or inflammation
* Injuries that to the decision of the provider of care, needs a targeted local treatment other than as provided for in the Protocol
* Patient / lesion that has already been previously recruited into the study, before a period of 10 days (wash-out) of suspension from the same research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | 1 month
Patient's pain | 1 month

SECONDARY OUTCOMES:
Clinical evaluation of the lesion scores for each visit | 1 month
The presence / absence of infection for each visit | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Bianchi, Study Director — Associazione Infermieristica per lo studio delle Lesioni Cutanee
Locations (1):
- Ospedale Bellaria - UOC Dermatologia, Bologna, Bologna, Italy